CLINICAL TRIAL: NCT04423913
Title: Evaluation of the Safety, Tolerability, Distribution and Dose Effect of Neoadjuvant Transarterial Chemoembolization With Doxorubicin in Prostate Cancer Patients at a High Risk of Recurrence Before Radical Prostatectomy: A Phase IIa Study
Brief Title: Safety, Tolerability, Distribution & Dose Effect of Neoadjuvant Transarterial Chemoembolization With Doxorubicin in Prostate Cancer Patients Before Radical Prostatectomy
Acronym: CAPEMCHAR
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NIMAO/2018-01/JF-01; 2019-001920-36 (EudraCT Number); 2019-A02946-51 (Registry Identifier: RCB No.)
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Prostate Cancer
Keywords: doxorubicin; beads; embolization; chemoembolization; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a purely descriptive, non randomized, non controlled, prospective sequential-type pilot study on the first use in the indication for prostatic arterial embolization using beads loaded with doxorubicin in increasing doses: 0 mg, 2.5mg, 5 mg and 10 mg. It is a study with escalating doses of doxorubicin : 3 patients with non-loaded beads, 3 patients with beads loaded at 2.5 mg (1/20 of the dose administered for liver tumors), 3 patients with beads loaded at 5mg and 3 patients with beads loaded at 10mg.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients undergoing transarterial embolization of the prostate (Experimental): Three patients will undergo transarterial embolization of the prostate using unloaded beads.
  Interventions: Other: Administration of embolization beads
- Transarterial prostatic chemoembolization, 2.5 mg doxorubicin (Experimental): Three patients will undergo transarterial chemoembolization of the prostate using beads loaded with 2.5 mg of doxorubicin.
  Interventions: Other: Administration of embolization beads
- Transarterial prostatic chemoembolization, 5.0 mg doxorubicin (Experimental): Three patients will undergo transarterial chemoembolization of the prostate using beads loaded with 5.0 mg of doxorubicin.
  Interventions: Other: Administration of embolization beads
- Transarterial prostatic chemoembolization, 10.0 mg doxorubicin (Experimental): Three patients will undergo transarterial chemoembolization of the prostate using beads loaded with 10.0 mg of doxorubicin.
  Interventions: Other: Administration of embolization beads

INTERVENTIONS:
Other: Administration of embolization beads — Patients will receive embolization beads, loaded with doxorubicin or not.

SUMMARY:
Our hypothesis is that the doxorubicin eluting-beads currently used in hepato-oncology might be applicable to high-grade prostate cancer before radical prostatectomy.

The primary objective of this Phase IIa pilot study is to evaluate the safety of performing prostate embolization with doxorubicin eluting-beads according to different loading doses. Four dose levels will be tested: doxorubicin-free beads to test the effect of embolization alone, 2.5 mg of doxorubicin (1/20 of the dose administered for liver cancers), 5 mg and 10 mg of doxorubicin.

The secondary objectives of the study are to evaluate the tolerance (functionnal questionaries at D0, D14 M1 and M3; collection of complications at D1, D5, D14, M1, M3; MRI at D14), evaluate the systemic diffusion of doxorubicin (doxorubinemia at D1), evaluate an early anti-tumor effect of the treatment (via a prostate-specific antigen test at D14 M1, M3 and magnetic resonance imaging at D14), describe the distribution of beads observed on the surgical specimen and evaluate the dose effect at 1 month and 3 months after surgery (via a prostate-specific antigen test at D14, M1, M3 and magnetic resonance imaging at D14).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given written informed consent.
* Patients must be affiliated to or benefit from a health insurance scheme.
* Patients with a high-risk prostate cancer with a Gleason score of 9-10 on the biopsy, candidate for a multimodal treatment with radical prostatectomy validated at the multidisciplinary meeting.
* Patients with a normal blood count.
* Patients with a normal liver function test.
* Patients with an electrocardiogram including left ventricle ejection fraction (ventricular scintigraphy or echocardiography) and an echocardiogram allowing us to rule out heart disease.
* Patient must be completely recovered from acute toxicities (such as stomatitis, neutropenia, thrombopenia and generalized infections) caused by a previous cytotoxic treatment.
* OMS/ECOG score≤1 (to guard against a possible loss of therapeutic opportunity related to a delay in surgery caused by chemo-embolization).

Exclusion Criteria:

* Patients who are taking part in another study.
* Patients in an exclusion period determined by a previous study.
* Patients under legal guardianship, curatorship or tutorship.
* Patients not in condition to be able to express his consent (e.g. patient undergoing psychiatric treatment with mental disorders)
* Patients who refuse to sign the consent form.
* Patients for whom it is impossible to give clear information. • Patient already has a metastatic disease.
* Patients who have contraindications for surgery.
* Patients with a rectal or vesicular collateral pathology that cannot be excluded or a collateral penile pathology which, by precaution, would not allow embolization (unknown effect on the erection in the event of arterial exclusion).
* Patients with a contraindication for magnetic resonance imaging (pacemaker incompatible with MRI, claustrophobia, metal apparatus, total hip prosthesis).
* Patients with a past history of aortobifemoral bypass procedure or other vascular surgery making endovascular access to the prostate arteries impossible.
* Patients with irreversible hemostasis disorder: TP < 50%, TCA > twice the control, Platelets < 60 G/L.
* Patients with contraindications as mentioned in the Summary of Product Characteristics for Doxorubicin.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As the study relates to embolization of prostate cancer, only male patients are concerned.
Enrollment: 12 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety of prostate embolization using unloaded beads. | Day 0 (i.e. on the day of the intervention)
  The number of serious undesirable events will be noted during the embolization. The undesirable event noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using unloaded beads. | Day 1 (i.e. one day after the intervention)
  The number of serious undesirable events will be noted the day after embolization. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using unloaded beads. | Day 5 (i.e. 5 days after the intervention)
  The number of serious undesirable events will be noted by telephone. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using unloaded beads. | Day 14 (i.e. 2 weeks after the intervention)
  This will be evaluated by magnetic resonance imaging (vesicular or rectal necrosis, fistula or abcess) and at the time of surgery.The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using unloaded beads. | Day 30 (i.e. 1 month after the intervention)
  Evaluation of post-operative complications. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using unloaded beads. | Three months after the intervention
  Evaluation of post-operative complications. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 2.5 mg of doxorubicin | Day 0 (i.e. on the day of the intervention)
  The number of serious undesirable events will be noted during the embolization. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 2.5 mg of doxorubicin | Day 1 (i.e. one day after the intervention)
  The number of serious undesirable events will be noted after the embolization. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 2.5 mg of doxorubicin | Day 5 (i.e. 5 days after the intervention)
  The number of serious undesirable events will be noted by telephone. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 2.5 mg of doxorubicin | Day 14 (i.e. 2 weeks after the intervention)
  This will be evaluated by magnetic resonance imaging (vesicular or rectal necrosis, fistula or abcess) and at the time of surgery.The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 2.5 mg of doxorubicin | Day 30 (i.e. 1 month after the intervention)
  Postoperative complications. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 2.5 mg of doxorubicin | Three months after the intervention
  Postoperative complications. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 5.0 mg of doxorubicin | Day 0 (i.e. on the day of the intervention)
  The number of serious undesirable events will be noted during the embolization. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 5.0 mg of doxorubicin | Day 1 (i.e. one day after the intervention)
  The number of serious undesirable events will be noted after the embolization. The side effects noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 5.0 mg of doxorubicin | Day 5 (i.e. 5 days after the intervention)
  The number of serious undesirable events will be noted by telephone. The undesirable events noted will be: intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 5.0 mg of doxorubicin | Day 14 (i.e. 2 weeks after the intervention)
  This will be evaluated by magnetic resonance imaging (vesicular or rectal necrosis, fistula, abcess) and at the time of surgery.The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 5.0 mg of doxorubicin | Day 30 (i.e. 1 month after the intervention)
  Postoperative complications. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 5.0 mg of doxorubicin | 3 months after the intervention
  Postoperative complications. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 10.0 mg of doxorubicin | Day 0 (i.e. on the day of the intervention)
  The number of serious undesirable events will be noted during the embolization. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 10.0 mg of doxorubicin | Day 1 (i.e. one day after the intervention)
  The number of serious undesirable events will be noted after the clinical embolization. The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 10.0 mg of doxorubicin | Day 5 (i.e. 5 days after the intervention)
  The number of serious undesirable events will be noted by telephone. The undesirable events noted will be: intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 10.0 mg of doxorubicin | Day 14 (i.e. 2 weeks after the intervention)
  This will be evaluated by magnetic resonance imaging (vesicular or rectal necrosis, fistula, abcess) and at the time of surgery.The undesirable events noted will be: non-targeted necrosis, intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 10.0 mg of doxorubicin | Day 30 (i.e. 1 month after the intervention)
  Postoperative complications. The undesirable events noted will be: intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.
Evaluation of safety of prostate embolization using beads loaded with 10.0 mg of doxorubicin | Three months after the intervention
  Postoperative complications. The undesirable events noted will be: intense vesicle or rectal pain, rectal bleeding, abundant hematuria and fever.

SECONDARY OUTCOMES:
Tolerance of prostate embolization using unloaded beads. | Day 14
  Dynamic contrast-enhanced Magnetic Resonance Imaging (1.5 or 3 Tesla multiparametric acquisition with T2 morphologic sequencing) will be performed to evaluate modifications in tumor volume and necrosis area.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin. | Day 14
  Dynamic contrast-enhanced Magnetic Resonance Imaging (1.5 or 3 Tesla multiparametric acquisition with T2 morphologic sequencing) will be performed to evaluate modifications in tumor volume and necrosis area.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin. | Day 14
  Dynamic contrast-enhanced Magnetic Resonance Imaging (1.5 or 3 Tesla multiparametric acquisition with T2 morphologic sequencing) will be performed to evaluate modifications in tumor volume and necrosis area.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin. | Day 14
  Dynamic contrast-enhanced Magnetic Resonance Imaging (1.5 or 3 Tesla multiparametric acquisition with T2 morphologic sequencing) will be performed to evaluate modifications in tumor volume and necrosis area.
Tolerance of prostate embolization using unloaded beads: Clavien-Dindo score | Day 14
  Postoperative complications evaluated according to the Clavien-Dindo score: bruising, arterial wound with bleeding, vesicle wound, rectal wound, parietal abcess, deep abcess…
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin:Clavien-Dindo score | Day 14
  Postoperative complications evaluated according to the Clavien-Dindo score: bruising, arterial wound with bleeding, vesicle wound, rectal wound, parietal abcess, deep abcess…
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin: Clavien-Dindo score | Day 14
  Postoperative complications evaluated according to the Clavien-Dindo score: bruising, arterial wound with bleeding, vesicle wound, rectal wound, parietal abcess, deep abcess…
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin: Clavien-Dindo score | Day 14
  Postoperative complications evaluated according to the Clavien-Dindo score: bruising, arterial wound with bleeding, vesicle wound, rectal wound, parietal abcess, deep abcess…
Tolerance of prostate embolization using unloaded beads : International Prostate Symptom Score | Day 14
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using unloaded beads : International Prostate Symptom Score | Day 30 (i.e. one month after embolization)
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using unloaded beads : International Prostate Symptom Score | Three months after embolization
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Evaluation of tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin : International Prostate Symptom Score | Day 14
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Evaluation of tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin : International Prostate Symptom Score | Day 30 (i.e. 1 month after embolization)
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Evaluation of tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin : International Prostate Symptom Score | Three months after embolization
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin : International Prostate Symptom Score | Day 14
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin : International Prostate Symptom Score | Day 30 i.e. 1 month after embolization
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin : International Prostate Symptom Score | Three months after embolization
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin : International Prostate Symptom Score | Day 14
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin : International Prostate Symptom Score | Day 30 (i.e. 1 month after embolization)
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin : International Prostate Symptom Score | Three months after embolization
  The International Prostate Symptom Score (IPSS) can be utilized to measure the severity of lower urinary tract symptoms. It is a validated, reproducible scoring system to assess disease severity and response to therapy. The IPSS is made up of 7 questions related to voiding symptoms. A score of 0 to 7 indicates mild symptoms, 8 to 19 indicates moderate symptoms and 20 to 35 indicates severe symptoms.
Tolerance of prostate embolization using unloaded beads : IIEF-6 score | Day 14
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using unloaded beads : IIEF-6 score | Day 30 (i.e. 1 month after embolization)
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using unloaded beads : IIEF-6 score | Three months after embolization
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin: IIEF-6 score | Day 14
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin: IIEF-6 score | Day 30 (i.e. one month after embolization)
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin: IIEF-6 score | Three months after embolization)
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin: IIEF-6 score | Day 14
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin: IIEF-6 score | Day 30 (i.e. 1 month after embolization)
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin: IIEF-6 score | Three months after embolization
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin: IIEF-6 score | Day 14
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin: IIEF-6 score | Day 30 (i.e.1 month after embolization)
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin: IIEF-6 score | Three months after embolization
  The International Index of Erectile Function (IIEF-6 ) score was developed and validated in 96-97 by Pfizer then adopted by the WHO as the gold standard for judging the efficacy of treatment for erection difficulties evaluated as part of clinical trials. It is the most commonly-used validated, multidimensional, self-administered questionnaire to evaluate erection difficulties (Rosen, Althof & Giuliano 2006). It consists of 15 questions covering 5 areas: erectile function (questions 1, 2, 3, 4, 5 and 15),satisfaction regarding sexual activity (questions 6,7 and 8), orgasm (questions 9 and 10), sexual desire (questions 11 and 12), overall satisfaction (questions 13 and 14). Patients must respond to the questionnaire based on their own experience over the last 4 weeks.
Tolerance of prostate embolization using unloaded beads : EORTC - QLQ-C30 score | Day 14
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using unloaded beads : EORTC - QLQ-C30 score | Day 30 (i.e. 1 month after embolization)
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using unloaded beads : EORTC - QLQ-C30 score | Three months after embolization
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin : EORTC - QLQ-C30 score | Day 14
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin : EORTC - QLQ-C30 score | Day 30 (i.e. 1 month after embolization)
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicin : EORTC - QLQ-C30 score | Three months after embolization
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin : EORTC - QLQ-C30 score | Day 14
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin : EORTC - QLQ-C30 score | Day 30 (i.e. 1 month after embolization)
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicin : EORTC - QLQ-C30 score | Three months after embolization
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin : EORTC - QLQ-C30 score | Day 14
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin : EORTC - QLQ-C30 score | Day 30 (i.e. 1 month after embolization)
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicin : EORTC - QLQ-C30 score | Three months after embolization
  The European Organisation for Research and Treatment of Cancer (EORTC) developed the QLQ-C30 self-questionnaire to evaluate the patient's quality of life after the intervention. It contains 28 questions with 4 possibilities of answers each with 4 possibilities: 1 = Not at All 2 = A Little 3 = Quite a Bit 4 = Very Much and two questions each with a seven-point Lickert scale in which 1 = very poor and 7 = excellent relating respectively to how the patient would rate his general health in the past week and how he would rate his quality of life in the past week.
Tolerance of prostate embolization using unloaded beads : 24h pad test | Day 14
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using unloaded beads : 24h pad test | Day 30 (i.e. 1 month after embolization)
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using unloaded beads : 24h pad test | Three months after embolization
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicine : 24h pad-test | Day 14
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicine : 24h pad-test | Day 30 (1 month after embolization)
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 2.5 mg of doxorubicine : 24h pad-test | Three months after embolization)
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicine : 24h pad test | Day 14
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicine : 24h pad test | Day 30 (i.e. 1 month after embolization)
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 5.0 mg of doxorubicine : 24h pad test | Three months after embolization
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicine : 24h pad test | Day 14
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicine : 24h pad test | Day 30 (1 month after embolization)
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Tolerance of prostate embolization using beads loaded with 10.0 mg of doxorubicine : 24h pad test | Three months after embolization
  The 24h pad-test, or incontinence test, is a way of objectively, qualitatively and quantitatively measuring urine leakage under trial conditions. The time limit is 24 hours. The weight of dry pads is compared with the weight of all wet pads after 24 hours.
Prostate-specific antigen level in patients treated with unloaded beads. | Day 14 before surgery
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with unloaded beads. | Day 30 (i.e. 1 month after embolization)
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with unloaded beads. | Three months after embolization
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 2.5 mg of doxorubicine . | Day 14 before surgery
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 2.5 mg of doxorubicine . | Day 30 (i.e. 1 month after embolization)
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 2.5 mg of doxorubicine . | Three months after embolization
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 5.0 mg of doxorubicine . | Day 14 before surgery
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 5.0 mg of doxorubicine . | Day 30 (i.e. month after embolization)
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 5.0 mg of doxorubicine . | Three months after embolization
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 10.0 mg of doxorubicine . | Day 14
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 10.0 mg of doxorubicine . | Day 30 (i.e. 1 month after embolization)
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Prostate-specific antigen level in patients treated with beads loaded with 10.0 mg of doxorubicine . | Three months after embolization
  This test measures the amount of prostate-specific antigen (PSA) in the patient's blood. PSA is a protein produced by both cancerous and noncancerous tissue in the prostate. It is useful for the early detection of cancer.
Biological checkup for patients treated with beads loaded with 2.5 mg of doxorubicine | Three months after embolization
  The following levels will be tested : uric acid, potassium, creatinin, calcium. phosphate)
Biological checkup for patients treated with beads loaded with 5.0 mg of doxorubicine | Three months after embolization
  The following levels will be tested : uric acid, potassium, creatinin, calcium.
Biological checkup for patients treated with beads loaded with 10.0 mg of doxorubicine | Three months after embolization
  The following levels will be tested : uric acid, potassium, creatinin, calcium.
Complete blood count for patients treated with beads loaded with 2.5 mg of doxorubicine | Three months after embolization
  The volume of hemoglobine, red blood cells, white blood cells, neutrophils, granulocytes,lymphocytes, monocytes, eosinophils, basophils and platelets will be measured platelets according to the traditional means.
Complete blood count for patients treated with beads loaded with 5.0 mg of doxorubicine | Three months after embolization
  The volume of hemoglobine, red blood cells, white blood cells, neutrophils, granulocytes,lymphocytes, monocytes, eosinophils, basophils and platelets will be measured platelets according to the traditional means.
Complete blood count for patients treated with beads loaded with 10.0 mg of doxorubicine | Three months after embolization
  The volume of hemoglobine, red blood cells, white blood cells, neutrophils, granulocytes,lymphocytes, monocytes, eosinophils, basophils and platelets will be measured platelets according to the traditional means.
Liver test for patients treated with beads loaded with 2.5 mg of doxorubicine | Three months after embolization
  The following elements will be measured and compared with the test results before treatment :
  * Aspartate aminotransaminase (ASAT), alanine aminotransferase (ALAT)
  * bilirubin
Liver test for patients treated with beads loaded with 5.0 mg of doxorubicine | Three months after embolization
  The following elements will be measured and compared with the test results before treatment :
  * Aspartate aminotransaminase (ASAT), alanine aminotransferase (ALAT)
  * bilirubin
Liver test for patients treated with beads loaded with 10.0 mg of doxorubicine | Three months after embolization
  The following elements will be measured and compared with the test results before treatment :
  * Aspartate aminotransaminase (ASAT), alanine aminotransferase (ALAT)
  * bilirubin
Cardiac ultrasound and electrocardiogram for patients treated with beads loaded with 2.5 mg of doxorubicine | Three months after embolization
  The left ventricular ejection fraction will be calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume).
Cardiac ultrasound and electrocardiogram for patients treated with beads loaded with 5.0 mg of doxorubicine | Three months after embolization
  The left ventricular ejection fraction will be calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume).
Cardiac ultrasound and electrocardiogram for patients treated with beads loaded with 10.0 mg of doxorubicine | Three months after embolization
  The left ventricular ejection fraction will be calculated by dividing the volume of blood pumped from the left ventricle per beat (stroke volume) by the volume of blood collected in the left ventricle at the end of diastolic filling (end-diastolic volume).
Systemic dosage of free doxorubicin in blood in patients treated with beads loaded with 2.5 mg of doxorubicine | Day 1
  A blood sample will be taken and the concentration of doxorubicin will be measured in mg/m2

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — CHU de Nîmes, Place du Professeur Debré, 30029 Nîmes Cedex
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France